CLINICAL TRIAL: NCT00919646
Title: Arrhythmia Detection With Adherent Patient Monitoring Study
Brief Title: Monitoring Arrhythmia Patients in in Hospital Monitoring
Acronym: ADAM
Status: Completed | Type: Observational
Sponsor: Corventis, Inc. (Industry)
Responsible Party: Madhuri Bhat, VP Regulatory and Clinical affairs, Corventis
Other Study IDs: COR-2009-001
Record Dates: First submitted 2009-06-10; First posted 2009-06-12 (Estimated); Last update posted 2010-02-04 (Estimated); Status verified 2010-02

CONDITIONS: Arrhythmias
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a prospective, single center, non-randomized study to evaluate the arrhythmia monitoring performance of the AVIVO™ System in a hospital setting.

DETAILED DESCRIPTION:
The AVIVO™ System will continuously monitor the patient's cardiac activity which will be compared to the performance of standard telemetry system.

ELIGIBILITY:
Inclusion Criteria:

* Is female or male, 18 years of age or older
* Undergoing in-hospital electrocardiographic monitoring for primarily cardiac reasons

Exclusion Criteria:

* Is participating in another clinical study that may confound the results of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Telemetry ward
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2009-04; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Imad Libbus, PhD, Study Director — Corventis, Inc.